CLINICAL TRIAL: NCT02205619
Title: Remaining Root Substance Comparing a New Ultrasonic Scaling Device, Hand Instrumentation and Subgingival Air Polishing With Glycine. An in Vivo and in Vitro Study
Brief Title: Amount of Cementum After Scaling, Root Planing and Glycine Air Polishing
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Dr.Esra Bozbay, PhD Student, University of Roma La Sapienza
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ABT-1233-RV
Record Dates: First submitted 2014-07-24; First posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Dental Diseases
Keywords: Residual cementum; root surface instrumentation; ultrasonic scaling; air polishing with glycine
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ultrasonic instrumentation (Experimental): Prior to extraction, the teeth (N = 12) were randomly included into ultrasonic instrumentation (Air Flow Master Piezon®, EMS SA, Nyon - Swiss) treatment group
  Interventions: Device: Air Flow Master Piezon®, EMS SA, Nyon, Swiss
- Hand instrumentation (Experimental): Prior to extraction, the teeth (N = 12) were randomly included into hand curette (Gracey curettes, American Eagle, Missoula, MT, USA) treatment group hand instrumentation (Gracey curettes 5/6, 11/12, 13/14 American Eagle, Missoula, MT, USA)
  Interventions: Device: Gracey curettes, American Eagle, Missoula, MT, USA
- subgingival airpolishing with glycine (Experimental): Prior to extraction, the teeth (N = 12) were randomly included into air-polishing (Air Flow Master Piezon®, EMS SA, Nyon - Swiss) with the glycine powder (Air-flow® Powder Perio, EMS) treatment group.
  subgingival airpolishing with glycine(Air-flow® Powder Perio, EMS SA, Nyon, Swiss)
  Interventions: Device: Air-flow® Powder Perio, EMS SA, Nyon, Swiss
- ultrasonic following airpolishing (Experimental): Prior to extraction, the teeth (N = 12) were randomly included into ultrasonic following airpolishing ( Air Flow Master Piezon®, EMS SA, Nyon, Swiss) (Air-flow® Powder Perio, EMS SA, Nyon, Swiss) with the glycine powder treatment group
  Interventions: Device: Air Flow Master Piezon®, EMS SA, Nyon, Swiss; Device: Air-flow® Powder Perio, EMS SA, Nyon, Swiss

INTERVENTIONS:
Device: Air Flow Master Piezon®, EMS SA, Nyon, Swiss — comparison of different instruments on root cementum: Instrumentations with US devices ( Air Flow Master Piezon®, EMS SA, Nyon, Swiss) were performed with medium power settings and with the use of water cooling (as instructed by the manufacturer). One approximal root surface (distal and mesial) of each tooth was randomly subjected to debridement and the other approximal surface was used as control. All the instrumentations of teeth were performed by a single operator. The criteria for adequate treatment were smooth, hard root surfaces, with no remnants of calculus. The cleanliness and smoothness of the root surface were checked using a fine dental explorer. The instrumentations were done under local anesthesia.
  Other Names: Piezoelectric ultrasonic instrumentation
  Arms: Ultrasonic instrumentation; ultrasonic following airpolishing
Device: Gracey curettes, American Eagle, Missoula, MT, USA — comparison of different instruments on root cementum Hand instruments (Gracey curettes 5/6, 11/12, 13/14 American Eagle, Missoula, MT, USA) were used for subgingival root instrumentation. The criteria for adequate treatment were smooth, hard root surfaces, with no remnants of calculus. The cleanliness and smoothness of the root surface were checked using a fine dental explorer. The instrumentations were done under local anesthesia.
  Other Names: hand instrumentation
  Arms: Hand instrumentation
Device: Air-flow® Powder Perio, EMS SA, Nyon, Swiss — comparison of different instruments on root cementum: Instrumentations with air polishing (Air-flow® Powder Perio, EMS SA, Nyon, Swiss) were performed with a special nozzle and medium power settings and with the use of water cooling (as instructed by the manufacturer). One approximal root surface (distal and mesial) of each tooth was randomly subjected to debridement and the other approximal surface was used as control. All the measurements and instrumentations of teeth were performed by a single operator. The criteria for adequate treatment were smooth, hard root surfaces, with no remnants of calculus. The cleanliness and smoothness of the root surface were checked using a fine dental explorer. The instrumentations were done under local anesthesia
  Other Names: subgingival airpolishing with glycine
  Arms: subgingival airpolishing with glycine; ultrasonic following airpolishing

SUMMARY:
The purpose of this study was to evaluate the residual cementum with the histological measurements and root surface topography with SEM evaluation using four periodontal treatment methods.

DETAILED DESCRIPTION:
Cementum is a component of the periodontium, and its major role is to serve as the site of attachment for principal collagen fibers (Sharpey' s fibers). In particular, cementum, by virtue of its structural and dynamic qualities, provides tooth attachment and maintenance of occlusal relationships between the jaws. Its multiple functions are fulfilled by the biological activity and reactivity of cementoblasts, which deposits two collagen-containing varieties of cementum with completely different properties. Periodontal disease is the local inflammation of the supporting tissues of teeth, it causes destruction of gingival tissues, bone loss and loss of connective tissue attachment to cementum. Since the relationship between local bacteria and periodontal disease has been proved and widely recognised, it is generally accepted that removal of pathogenic microorganisms that form plaque and calculus is the major goal of periodontal treatment. This therapy currently consists of scaling and root planing, but in addition to mechanical instrumentation, regeneration and restoration of various periodontal components to their original form, function and consistency should be performed.

Previously it was accepted that bacterial endotoxins or bacteria penetrate the cementum of periodontally diseased root surfaces. Therefore, besides the removal of the subgingival plaque and calculus deposits, the removal of all or most of the cementum was one of the primary endpoints of periodontal healing. The goal of periodontal therapy was to attain a planed root surface with a smooth and hard surface characteristics and free of endotoxins as the cementum of a tooth prior to eruption. While some studies have reported that endotoxins are not located within cementum it has been accepted that the removal of 'diseased' cementum was not necessary for a successful periodontal treatment.

Saygin et al. reported that cementum is the site where soft-tissue attachment has to be re-established, and cementum matrix is a rich source of many growth factors which influence the activities of various periodontal cell types and Grzesik et al. stated that cementum plays a regulatory role in periodontal regeneration. From these studies it can be concluded that non-aggressive periodontal treatment is necessary for optimal periodontal health as well as for periodontal regeneration.

During periodontal therapy subgingival instrumentation by means of the removal of root cementum can be eventually lead to exposure of dentinal tubules, pulp injury and dentin hypersensitivity. The in vitro studies including establishing in vitro experimental models under standardized experimental conditions evaluated the amount of cementum with various instruments or force combinations. Several studies, which showed the effects of different instruments on root surfaces, emphasized that periodontal treatment can be performed less aggressively with respect to the removal of cementum.

Previously reported that the teeth treated by HC and US can present a surface without cementum and the open dentinal tubules.They reported that root surfaces treated by US showed a scaly and rough topography whether the teeth treated with HC presented smooth surfaces. Kawashima and co-workers compared two different piezoelectric US (VectorTM and EnacR scaler) and HC and found that both US groups had significantly more remaining cementum than the HC group. However they observed some areas with thin or absent cementum in the HC group. Ruhling et al. compared the effects of the piezoelectric US, sonic scaler (SS), sonic scaler insert coated with Teflon tube, Periotor insert and HC. They showed that HC and SS group presented greater removal of root cementum and nearly all cementum was removed in 25% of the samples treated with HC.

Tomasi et al. reported that biofilm and calculus certainly should be removed but also they questioned the requirement for removal of contaminated root cementum by root planing. US with new shaped tips and AP devices as alternative to HC designed for subgingival access have been developed for minimal root damage. In recent years, there are newly developed instruments presenting clinically efficient results in the treatment of chronic periodontitis. Subgingival AP has been suggested as a treatment modality for root debridement. Two recent studies have investigated the clinical and microbiological efficacy of subgingival AP by glycine powder in periodontal pockets and they revealed probing depth reductions and removal of subgingival biofilm. Today there is no scientific research evidence showing the loss of root substance or surface roughness by subgingival AP or US instrumentation with AP.

The aim of the present study was to compare the effect of in vivo root instrumentation using a new piezoelectric US instrument, HC and air polishing by glycine powder, under routine clinical conditions, on the thickness and surface characteristics of cementum.

Forty-eight periodontally involved caries free, single rooted teeth with advanced periodontitis scheduled for extraction treated in four different methods. The teeth were instrumented subgingivally at one approximal site either by hand curettes (HC), piezoelectric ultrasonic scaler (US), piezoelectric ultrasonic scaler following air polishing, air polishing (AP) alone. Upon extracting the teeth, instrumented and other non-instrumented sites analyzed with a dissecting microscope and SEM for the measurement of amount and surface characteristics of residual cementum.

ELIGIBILITY:
Inclusion Criteria:

* systemic factors (no systemic diseases; no medications affecting periodontal status in the previous 6 months; no pregnancy or lactation;
* behavioral factors (no smoking habits);
* dental and periodontal factors not to have had previous periodontal therapy; no class III dental mobility;
* a periodontal probing depth (PPD) ≥ 4 mm in at least two sites per tooth with single rooted ;
* have no caries or restorations on the mesial and distal surfaces and bleeding on probing.

Exclusion Criteria:

* systemic diseases; medications affecting periodontal status in the previous 6 months; pregnancy or lactation
* smoking habits
* have caries or restorations on the mesial and distal surfaces and bleeding on probing.
* have had previous periodontal therapy; class III dental mobility;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
thickness of cementum | within the first 60 days after extractions
  After instrumentations the teeth extractions (n=48) were done and the teeth were stored in the solution of NaCl. Upon extracting the teeth were sectioned perpendicularly to the root axis with a microtome (Leica, RM2245, Wetzlar, Germany) between 10 and 15 µm thickness and stained with hematoxylin and eosin (Leica Autostainer XL, Wetzlar, Germany). Two horizontally root sections of each tooth were taken from coronal and apical part of instrumented area for a total 96 histologic specimens. Coronal sections were taken 1 mm apically from the gingival margin, whereas apical sections were taken 1 mm coronally from the endpoint of periodontal pocket. The teeth were examined by an optic microscope (Nikon Eclipse i5, Tokyo, Japan) connected to a camera (Nikon, DS-Filc, Tokyo, Japan) and finally to a dedicated computer. The thickness of the cementum was measured by a specific software (Nikon, NIS Elements 4.0, Tokyo, Japan).

SECONDARY OUTCOMES:
Remaining calculus index (RCI) with SEM evaluation | within 30 days after extractions
  Before sectioning, the root surface characteristics of 20 randomly selected teeth were analyzed under scanning electron microscopy (LEO, EO 435 VP, Marvell Nanofabrication, Berkeley, CA, USA). The roots were gold-sputtered with a sputtering device (Agar Sputter Coater, 108 Supply 230, Frequency 50, Essex, UK). Micrographs were taken at magnifications from x48 to x210. Remaining calculus index (RCI) were scored as:0: No calculus remaining on the root surface 1: Small patches of extraneous material, probably consisting of calculus 2: Definite patches of calculus confined to relatively small areas 3: Considerable amount of remaining calculus, appearing as one or a few voluminous patches or as several smaller patches scattered on the treated surface.However, calculus appearance was provided with qualitative information on the mineral and organic composition of the root surface. Additionally, damages, scratches, gouges, cracks, cementum presence and changes in the cementum were noted.

OTHER OUTCOMES:
Roughness Loss of Tooth Substance Index (RLTSI) with SEM evaluation | within 30 days after teeth extractions
  Before sectioning, the root surface characteristics of 20 randomly selected teeth were analyzed under scanning electron microscopy (LEO, EO 435 VP, Marvell Nanofabrication, Berkeley, CA, USA). The roots were gold-sputtered with a sputtering device (Agar Sputter Coater, 108 Supply 230, Frequency 50, Essex, UK). Micrographs were taken at magnifications from x48 to x210. Roughness Loss of Tooth Substance Index (RLTSI) were scored as:0: Smooth or even root surface, without marks from the instrumentation and with no loss of tooth substance 1: Slightly roughened or corrugated local areas confined to the cementum 2: Definitely corrugated local areas where the cementum may be completely removed, although most of the cementum is still present 3: Considerable loss of tooth substance, with instrumentation marks extending into the dentin. The cementum is completely removed in large areas or there are a considerable number of lesions due to the instrumentation

CONTACTS AND LOCATIONS:
Overall Officials: Esra Bozbay, Dr, Principal Investigator — *Department of Dentistry and Maxillofacial Surgery, Section of Periodontics, School of Dentistry, Sapienza University of Rome, Rome, Italy.; Francesco Dominici, Dr, Study Chair — *Department of Dentistry and Maxillofacial Surgery, Section of Periodontics, School of Dentistry, Sapienza University of Rome, Rome, Italy.; Serdar Cintan, Prof, Study Chair — †Department of Periodontology, Faculty of Dentistry, Istanbul University, Istanbul, Turkey.; Aslan Yasar Gokbuget, Prof, Study Chair — †Department of Periodontology, Faculty of Dentistry, Istanbul University, Istanbul, Turkey.; Luigi Guida, Prof, Study Chair — ‡Department of Odontostomatological, Orthodontic and Surgical Disciplines, Second University of Naples, Naples, Italy.; Mehmet Serif Aydin, MSc Bio, Study Chair — §Department of Histology and Embryology, Faculty of Medicine, Bezmialem Vakif University, Istanbul, Turkey.; Andrea Pilloni, Prof, Study Director — *Department of Dentistry and Maxillofacial Surgery, Section of Periodontics, School of Dentistry, Sapienza University of Rome, Rome, Italy.